CLINICAL TRIAL: NCT03661840
Title: Acceptance and Commitment Therapy for Chronic Pain in Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-1102.cc
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Results first posted 2024-01-03 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Chronic Pain
Keywords: Acceptance and Commitment Therapy; Cancer; Survivor; Group Based; Pain Management
MeSH Terms: conditions — Chronic Pain; Neoplasms; Agnosia | interventions — Acceptance and Commitment Therapy; Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to the acceptance and commitment therapy intervention or to treatment as usual.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance and Commitment Therapy (Experimental): Participants will receive both the ACT intervention and medication management that is given as usual treatment.
  Interventions: Behavioral: Acceptance and Commitment Therapy
- Treatment as Usual (Active Comparator): Treatment as usual will include ongoing provision of usual treatment options for pain management.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — Intervention group participants will attend eight weekly, 90-minute, in person, group-based ACT sessions. Groups will be initiated with no more than 10 participants and no fewer than 6 participants. Sessions will include key theoretical ACT constructs and strategies as they relate to chronic pain. A licensed clinical psychologist or licensed clinical social worker trained in ACT will facilitate all sessions. Participants in the ACT intervention group will also continue to receive medication management and other behavioral management interventions that they would get as usual treatment.
  Arms: Acceptance and Commitment Therapy
Other: Treatment as Usual — Treatment as usual will include ongoing provision of usual treatment options for pain management. This includes continued medication management for cancer related chronic pain by prescribing providers, and access to supportive oncology services. It may also include other behavioral pain management such as physical therapy, acupuncture, or massage.
  Arms: Treatment as Usual

SUMMARY:
A study to help manage chronic pain in cancer survivors through Acceptance and Commitment Therapy (ACT) after undergoing active cancer treatment, such as surgery, chemotherapy, and/or radiation.

DETAILED DESCRIPTION:
This study attempts to apply effective pain management interventions from other chronic pain populations to those of cancer related populations. It will assess the ability of ACT to alleviate chronic cancer related pain and evaluate ease of implementation of treatment. Patients will be allocated to either the intervention group (ACT) or the control group, getting them the usual course of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Provision to sign and date the consent form
2. Stated willingness to comply with all study procedures and be available for the duration of the study
3. Be a male or female aged 18-100
4. Have pathology confirmed diagnosis of a solid tumor cancer
5. Be three or more months out from active cancer treatment (surgery, chemotherapy, and/or radiation)
6. Endorses experiencing pain for three or more months prior to eligibility screening
7. Indicates moderate to severe difficulties with pain interference as related to their cancer experience, with a score of 4 or higher on the pain interference item from the Chronic Pain Grading Questionnaire
8. Shows no evidence of cancer disease (NED) or with stable, chronic disease under "watchful waiting"
9. Fluent in English
10. Psychiatric stability as assessed by chart review and study personnel (e.g., not exhibiting symptoms consistent with diagnoses of serious mental illness such as active psychosis or mania)

Exclusion Criteria:

1. Having pain that can be solely attributed to a diagnosis outside of their cancer experience
2. Presenting with barriers to group participation (e.g., social anxiety) or when group-based provision of care would impede participant's treatment or that of other group members
3. Patients with a diagnosis of malignant neoplasm of the brain (ICD-10 C71) or malignant neoplasm of spinal cord, cranial nerves and other parts of central nervous system (ICD-10 C72).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elissa Kolva, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acceptance and Commitment Therapy | Treatment as Usual
Started | 28 | 22
Completed | 28 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acceptance and Commitment Therapy | Treatment as Usual | Total
Number analyzed (Participants) | 28 | 22 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 17 | 37
  >=65 years | 8 | 5 | 13
Age, Continuous [Mean (Full Range); unit: years] | 53 [31 to 75] | 56 [32 to 80] | 56 [31 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 17 | 40
  Male | 5 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 26 | 21 | 47
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 25 | 21 | 46
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 22 | 50

OUTCOME MEASURES:

1. Primary Outcome: The Degree of Effectiveness of Acceptance and Commitment Therapy: [Impact]
Description: Use the Medical Outcomes Study 36-Item Short Form Health Survey to assess physical health.
  Min = 0 Max = 100 Higher scores are better.
Time Frame: From baseline to 12 weeks post intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Intervention: Received acceptance and commitment therapy.
- Control: Treatment as usual
Arm/Group | Intervention | Control
Number analyzed (Participants) | 28 | 22
units on a scale
  Baseline | 23.9 (34.0) | 21.4 (29.9)
  12 week | 41.7 (39.9) | 37.5 (41.3)
Statistical Analysis 1: Comparison: Intervention vs Control; Sample size was estimated using d= 0.61, with power at 0.80 and α = .05, two-tailed. It is assumed that the correlation between pre and post-test measures will be high at .5. With these parameters and using repeated measures ANOVA to evaluate treatment difference, sample size is powered for clinical outcomes at 92 participants; with an estimated 30% attrition and conservatively including the possibility of screening failures, a maximum sample of 140 participants will be targeted for enrollment; Test type: Superiority; p = 0.82, Regression, Linear — Unadjusted model comparing the mean difference (change from 12 weeks - baseline) in outcome by intervention group; Mean Difference (Final Values) = 3.9, 95% CI 2-sided [-31 to 39], Standard Error of Mean 17

2. Primary Outcome: The Degree of Effectiveness of Acceptance and Commitment Therapy: [Impact]
Description: Use the Medical Outcomes Study 36-Item Short Form Health Survey to assess emotional wellbeing.
  Min=0 Max=100 Higher scores indicate better emotional wellbeing.
Time Frame: From baseline to 12 weeks post intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 28 | 22
units on a scale
  Baseline | 62.6 (18.3) | 74.1 (17.4)
  12-week follow up | 73.9 (14.5) | 72.9 (14.5)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.06, Regression, Linear — Unadjusted model comparing the change in outcome by intervention group; Mean Difference (Final Values) = 12, 95% CI 2-sided [-0.7 to 25], Standard Error of Mean 6.4
Statistical Analysis 2: Comparison: Intervention; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.05, ANOVA; Mean Difference (Final Values) = 0.61

3. Secondary Outcome: Number of Participants Who Want to Use Acceptance and Commitment Therapy as a Method for Treating Chronic Pain Post Active Cancer Treatment Active Cancer Treatment
Description: Feasibility of the intervention will be assessed through the collection of participant enrollment and adherence data throughout the intervention period and follow-up.
  We report the count of participants at each therapy session. Therapy sessions were held from baseline through week 8.
Time Frame: From baseline to end of intervention (weeks 1- 8)
Population: Data were only collected for the intervention group.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 28
Participants
  week1 therapy | 19
  week 2 therapy | 19
  week 3 therapy | 18
  week4 therapy | 18
  week5 therapy | 14
  week6 therapy | 18
  week7 therapy | 17
  week8 therapy | 17

4. Secondary Outcome: The Degree to Which Patients Enjoy Using Acceptance and Commitment Therapy as a Method for Treating Chronic Pain Post Active Cancer Treatment: [Acceptability]
Description: Acceptability of the intervention will be assessed through weekly ratings using a 5-point Likert scale for each session with intervention group members. The mean score is reported.
  Min = 1, Max = 5. Higher scores are better (i.e., indicate greater acceptability of the intervention).
Time Frame: From baseline to end of intervention (weeks 1- 8)
Population: Adherence was only collected for the intervention arm that received the therapy sessions.
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 28
units on a scale
  Week 1 | 4.4 [3 to 5]
  Week 2 | 4.5 [3 to 5]
  Week 3 | 4.6 [4 to 5]
  Week 4 | 4.6 [3 to 5]
  Week 5 | 4.6 [3 to 5]
  Week 6 | 4.6 [3 to 5]
  Week 7 | 4.8 [4 to 5]
  Week 8 | 4.8 [4 to 5]

5. Secondary Outcome: The Ability of Methodological Strategies Used to Monitor and Enhance the Reliability and Validity of ACT: [Fidelity]
Description: Fidelity of the treatment will be assessed through the use of a standardized checklist of core intervention components. It is measured as the mean percent of content checklist items presented to groups each week.
Time Frame: From baseline to end of intervention (weeks 1- 8)
Population: Limited to intervention group.
Measure: Mean (Standard Deviation); unit: percentage of content checklist items
Arm/Group | Intervention
Number analyzed (Participants) | 28
percentage of content checklist items
  Week 1 | 100 (0)
  Week 2 | 100 (0)
  Week 3 | 100 (0)
  Week 4 | 100 (0)
  Week 5 | 100 (0)
  Week 6 | 100 (0)
  Week 7 | 100 (0)
  Week 8 | 100 (0)

ADVERSE EVENTS:
Time Frame: Time from baseline to 12 week follow up.
Arm/Group | Acceptance and Commitment Therapy | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/22
Other Adverse Events (participants affected / at risk) | 0/28 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-03-30): https://cdn.clinicaltrials.gov/large-docs/40/NCT03661840/Prot_SAP_ICF_000.pdf